CLINICAL TRIAL: NCT05397470
Title: A Phase 3 Global, Randomized, Double-Blind, Placebo-Controlled, 48-Week, Parallel-Group Study of the Efficacy and Safety of Losmapimod in Treating Patients With Facioscapulohumeral Muscular Dystrophy (FSHD) (REACH)
Brief Title: Efficacy and Safety of Losmapimod in Treating Participants With Facioscapulohumeral Muscular Dystrophy (FSHD) (REACH)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Fulcrum Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1821-FSH-301
Record Dates: First submitted 2022-05-04; First posted 2022-05-31 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Facioscapulohumeral Muscular Dystrophy (FSHD)
Keywords: Facioscapulohumeral muscular dystrophy (FSHD); Facioscapulohumeral muscular dystrophy type 1 (FSHD 1); Facioscapulohumeral muscular dystrophy type 2 (FSHD 2); Muscular Dystrophy; Facioscapulohumeral Muscular Disorders; Musculoskeletal Diseases; Neuromuscular Diseases; REACH
MeSH Terms: conditions — Muscular Dystrophy, Facioscapulohumeral; Muscular Dystrophies; Musculoskeletal Diseases; Neuromuscular Diseases | interventions — 6-(5-((cyclopropylamino)carbonyl)-3-fluoro-2-methylphenyl)-N-(2,2-dimethylprpyl)-3-pyridinecarboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part B of the study will be performed in an open-label fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part A: Placebo-controlled treatment period: Losmapimod (Experimental): Participants will be randomized to receive losmapimod.
  Interventions: Drug: Losmapimod
- Part A: Placebo-controlled treatment period: Placebo (Placebo Comparator): Participants will be randomized to receive placebo
  Interventions: Drug: Placebo oral tablet
- Part B: Open-label extension (Experimental): Participants will receive losmapimod, upon completion of all assessments for Part A.
  Interventions: Drug: Losmapimod

INTERVENTIONS:
Drug: Losmapimod — Losmapimod 15 mg will be administered BID by mouth along with food.
  Arms: Part A: Placebo-controlled treatment period: Losmapimod; Part B: Open-label extension
Drug: Placebo oral tablet — Placebo will be administered BID by mouth along with food.
  Arms: Part A: Placebo-controlled treatment period: Placebo

SUMMARY:
This is a study to evaluate the safety and efficacy of losmapimod in treating participants with Facioscapulohumeral Muscular Dystrophy (FSHD). Participants diagnosed with Facioscapulohumeral muscular dystrophy type 1 (FSHD1) or Facioscapulohumeral muscular dystrophy type 2 (FSHD2) will participate in Part A (Placebo-controlled treatment period) and will be randomized in a 1:1 ratio to receive losmapimod 15 milligrams (mg) or placebo orally twice daily (BID). Upon completion of Part A, participants will have the option to rollover into Part B (open-label extension) to evaluate the long-term safety, tolerability, and efficacy of losmapimod and will receive losmapimod 15 mg orally BID.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants must be between 18 and 65 years of age, inclusive.
* Genetically confirmed diagnosis of FSHD 1 or FSHD 2.
* Clinical severity score of 2 to 4 (Ricci Score; Range 0-5), at screening. Participants who are wheelchair-dependent or dependent on walker or wheelchair for activities are not permitted to enroll in the study.
* Screening total RSA (Q1-Q4) without weight in the dominant UE assessed by RWS ≥ 0.2 and ≤ 0.7.
* No contraindications to MRI.

Key Exclusion Criteria:

* Previously diagnosed cancer that has not been in complete remission for at least 5 years. Localized carcinomas of the skin and carcinoma in situ of the cervix that have been resected or ablated for cure are not exclusionary.
* Participants who are on drug(s) or supplements that may affect muscle function, as determined by the Investigator: participants must be on a stable dose of that drug(s) or supplement for at least 3 months prior to the first dose of study drug and remain on that stable dose for the duration of the study.
* Known active opportunistic or life-threatening infections including Human Immunodeficiency virus (HIV) and hepatitis B or C.
* Known active or inactive tuberculosis infection.
* Acute or chronic history of liver disease.
* Known severe renal impairment.
* History of cardiac dysrhythmias requiring anti-arrhythmia treatment(s); or history or evidence of abnormal ECGs.
* Use of another investigational product within 30 days or 5 half-lives (whichever is longer) or currently participating in a study of an investigational device.
* Current or anticipated participation in a natural history study. Previous participation is allowed but participants cannot continue after enrollment in Study 1821-FSH-301.
* Known hypersensitivity to losmapimod or any of its excipients.
* Previous participation in a Fulcrum-sponsored FSHD losmapimod study (FIS-001-2019 or FIS-002-2019).

Note that all other inclusion and exclusion criteria are listed in the protocol and only key are presented.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2024-11-19 (Actual); Study Completion 2024-11-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (14):
  - University of California Irvine, Irvine, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Florida, Gainesville, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Rochester Medical Center, Rochester, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - Nice University Hospital - CHU Nice, Nice, PACA
  - Institute de Myologie, Groupe Hospitalier Pitié-Salpêtrière, Paris
- Germany (3):
  - University Hospital Bonn, Bonn
  - LMU Klinikum Ludwig-Maximilians-Universität München, München
  - Universitätsklinikum Ulm, Ulm
- Italy (2):
  - Fondazione Serena Onlus- Centro Clinico NEMO, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - Leiden University Medical Centre, Leiden, Southern Holland
- Spain (3):
  - Hospital Universitario Donostia, San Sebastián, Guipuzkoa
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - University College of London Hospitals, London
  - Newcastle upon Tyne NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of a manuscript describing the clinical trial data, Fulcrum will provide access to all collected, individual, de-identified participant data and related study documents (e.g., Study Protocol, Statistical Analysis Plan [SAP]) through a third party. Access will be granted upon request from qualified researchers and will be subject to specific criteria and conditions.
  Further details, including the IPD sharing URL, will be provided in an update to this posting.

REFERENCES:
- [Background] Barbour AM, Sarov-Blat L, Cai G, Fossler MJ, Sprecher DL, Graggaber J, McGeoch AT, Maison J, Cheriyan J. Safety, tolerability, pharmacokinetics and pharmacodynamics of losmapimod following a single intravenous or oral dose in healthy volunteers. Br J Clin Pharmacol. 2013 Jul;76(1):99-106. doi: 10.1111/bcp.12063. PMID 23215699
- [Background] Han JJ, Kurillo G, Abresch RT, de Bie E, Nicorici A, Bajcsy R. Reachable workspace in facioscapulohumeral muscular dystrophy (FSHD) by Kinect. Muscle Nerve. 2015 Feb;51(2):168-75. doi: 10.1002/mus.24287. Epub 2014 Nov 19. PMID 24828906
- [Background] Mellion ML, Ronco L, Berends CL, Pagan L, Brooks S, van Esdonk MJ, van Brummelen EMJ, Odueyungbo A, Thompson LA, Hage M, Badrising UA, Raines S, Tracewell WG, van Engelen B, Cadavid D, Groeneveld GJ. Phase 1 clinical trial of losmapimod in facioscapulohumeral dystrophy: Safety, tolerability, pharmacokinetics, and target engagement. Br J Clin Pharmacol. 2021 Dec;87(12):4658-4669. doi: 10.1111/bcp.14884. Epub 2021 May 14. PMID 33931884
- [Derived] Voermans NC, Statland JM, Hayward LJ, Rosenbohm A, Lopez de Munain A, Sacconi S, Leung DG, Badrising UA, Vissing J, Schoser B, Muelas N, Lochmuller H, Bugiardini E, Wang LH, Maggi L, Ragole T, Pestronk A, Hamel JI, Goyal NA, Korngut L, Naddaf E, Harper A, Shieh PB, Kornblum C, Sansone V, Genge A, Tasca G, Jiang J, Jouvin MH, Tawil R; REACH Investigators. A randomized, double-blind, placebo-controlled study of losmapimod in patients with facioscapulohumeral muscular dystrophy: Results of the REACH study. J Neuromuscul Dis. 2026 Feb 6:22143602261419558. doi: 10.1177/22143602261419558. Online ahead of print. PMID 41649965

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-part study. Part A was a global, randomized, double-blind, placebo-controlled, parallel-group, multicenter study that enrolled up to 260 participants. Part B was an open-label extension phase in which approximately 249 participants from Part A rolled over to receive Losmapimod treatment.
Pre-assignment Details: Participants who completed 48 Weeks treatment period in Part A were enrolled in Part B. Part A of the study was completed as planned; however, Part B was terminated prematurely due to a Sponsor decision.
Groups:
- Part A: Losmapimod 15 Milligrams (mg): Participants received Losmapimod 15 mg orally twice daily (BID) with food for 48 weeks.
- Part A: Placebo: Participants received matching placebo orally twice daily (BID) with food for 48 weeks.
- Part B: Losmapimod 15 mg OLE: Participants who completed Part A rolled over into Part B and received Losmapimod 15 mg orally twice daily (BID) with food.
Period: Part A: PCT Period (Up to 48 Weeks)
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo | Part B: Losmapimod 15 mg OLE
Started | 130 | 130 | 0
Completed | 127 | 126 | 0
Not Completed | 3 | 4 | 0
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Other | 0 | 1 | 0
Period: Part B: OLE Period (Up to Week 127)
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo | Part B: Losmapimod 15 mg OLE
Started | 0 | 0 | 249
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 249
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Study closed/terminated | 0 | 0 | 244

BASELINE CHARACTERISTICS:
Population: Full Analysis Set comprised of all participants with FSHD1 or FSHD2 who are randomized and receive at least 1 dose of study drug in the placebo-controlled treatment period.
Groups:
- Losmapimod 15 mg: Participants received Losmapimod 15 mg orally twice daily (BID) with food for 48 weeks.
- Matching Placebo: Participants received matching placebo orally twice daily (BID) with food for 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Losmapimod 15 mg | Matching Placebo | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (12.3) | 44.3 (12.0) | 43.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 59 | 115
  Male | 74 | 71 | 145
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 113 | 112 | 225
  Unknown or Not Reported | 9 | 12 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 115 | 116 | 231
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Total Relative Surface Area (RSA) Quadrants 1 to 5 (Q1-Q5) With 500 Grams (g) Wrist Weight Averaged Over Both Arms as Assessed by Reachable Workspace (RWS) at Week 48
Description: Participants are instructed to complete a simple set of standardized movements of each arm centered around the shoulder joint. These arm movements are captured and quantitated with the use of a video camera. The RWS is a clinical outcome measure that measures the relative surface area that a participant may reach with an outstretched arm. Responses are rated on a scale of 0 (no reachable workspace) to 1.25 (maximal reachable workspace). Higher scores indicate better outcomes. Baseline is the last non-missing evaluation prior to first dose of study drug. Change from Baseline was calculated as the post-treatment value minus the value at Baseline.
Time Frame: Baseline (Day 1) and at Week 48
Population: Full Analysis Set comprised of all participants with FSHD1 or FSHD2 who are randomized and receive at least 1 dose of study drug in the placebo-controlled treatment period. Only those participants with data available at specified timepoints has been presented.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 122 | 121
Scores on a scale | 0.013 (0.007) | 0.010 (0.007)
Statistical Analysis 1: Comparison: Part A: Losmapimod 15 Milligrams (mg) vs Part A: Placebo; Test type: Other; p = 0.7501, Mixed Model Repeated Measures; Least square mean difference = 0.003, 95% CI 2-sided [-0.014 to 0.020]

2. Primary Outcome: Part B: Number of Participants Reporting Serious Treatment Emergent Adverse Events (Serious TEAEs) and Non-serious TEAEs > 5%
Description: Treatment-emergent adverse event is an AE that begins on or after the first dose of study drug and on or before the stop of study drug + 35 days or begins before the first dose of study drug and worsens on or after the first dose of study drug and on or before the stop of study drug + 35 days. A SAE is defined as an AE that results in any of the following outcomes: death; life-threatening adverse event; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; congenital anomaly/birth defect.
Time Frame: Week 48 to Week 127
Population: Open-Label Analysis Set comprises of all participants who received at least 1 dose of losmapimod in Part B.
Measure: Count of Participants; unit: Participants
Groups:
- Part B: Open Label Treatment Period: Losmapimod: Participants who completed Part A rolled over into Part B and received Losmapimod 15 mg orally twice daily (BID) with food.
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants
  Any serious TEAE | 7
  Any non-serious TEAE > 5% | 94

3. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Chemistry Parameters
Description: Blood samples were collected for the analysis of chemistry parameters: Glucose, sodium, potassium, calcium, inorganic phosphate, total protein, albumin, blood urea nitrogen, creatinine, total bilirubin, direct bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, gamma glutamyl transferase and creatine phosphokinase.
Time Frame: Week 48 to Week 127
Population: Open-label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants | 0

4. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: Blood samples were collected for the analysis of hematology parameters: hemoglobin (including mean corpuscular volume), mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, hematocrit, red blood cell count, total white blood cell count, platelet count. Differential blood counts, including basophils, eosinophils, neutrophils, lymphocytes, and monocytes
Time Frame: Week 48 to Week 127
Population: Open-label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants | 0

5. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Urinalysis
Description: Urine samples were collected for the analysis of urinalysis parameters: Leucocytes, blood, nitrite, protein, urobilinogen, bilirubin, potential of Hydrogen (pH), specific gravity, ketones, glucose.
Time Frame: Week 48 to Week 127
Population: Open-label Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants | 0

6. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Vital Parameters
Description: Vital parameters including pulse rate, respiration rate, blood pressure, and temperature were measured in seated or recumbent for at least 5 minutes. Data for number of participants with abnormal clinically significant changes for vital signs have been presented.
Time Frame: Week 48 to Week 127
Population: Open-label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants | 0

7. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: Twelve-lead ECGs were performed after participants has been recumbent for at least 5 minutes.
Time Frame: Week 48 to Week 127
Population: Open-label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants | 0

8. Primary Outcome: Part B: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: Physical examinations included an evaluation of body systems, including but not limited to the following: skin; head, eyes, ears, nose, and throat; respiratory system; cardiovascular system; abdomen (liver, spleen); lymph nodes; neurological system; and musculoskeletal system.
Time Frame: Week 48 to Week 127
Population: Open-label Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Open Label Treatment Period: Losmapimod
Number analyzed (Participants) | 249
Participants | 0

9. Secondary Outcome: Part A: Change From Baseline in Quality of Life in Neurologic Disorders Upper Extremity (Neuro-QoL UE) Scale at Week 48
Description: The Neuro-QoL Upper Extremity (UE) scale is a patient-reported outcome measure designed to assess upper limb function in individuals with neurologic conditions. It evaluates a participant's self-reported difficulty in performing activities for daily living (ADLs) involving digital, manual, and reach-related function and self-care. Responses are divided into 5 ordinal levels (1 = unable to do, 2 = with much difficulty, 3 = with some difficulty, 4 = with a little difficulty, 5 = without any difficulty). Lower scores indicate worse symptoms. Change from Baseline was calculated as the post-treatment value minus the value at Baseline.
Time Frame: Baseline (Day 1) and at Week 48
Population: Full Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 120 | 125
Scores on a scale | -2.10 (3.82) | -1.51 (3.68)

10. Secondary Outcome: Part A: Number of Participants With Response to Patient's Global Impression of Change (PGIC) at Week 48
Description: The Patient Global Impression of Change (PGIC) is a standard participant-report outcome that measures the participant's self-reported change in health status compared to the start of the study. The PGIC uses a single question and 7-point patient self-reporting scale of overall improvement during treatment ranging from 1 (very much improved) to 7 (very much worse). Higher scores indicate worse symptoms.
Time Frame: At Week 48
Population: Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants
  Very much improved | 1 | 2
  Much improved | 7 | 5
  Minimally improved | 28 | 24
  No change | 43 | 47
  Minimally worse | 36 | 36
  Much worse | 10 | 12
  Very much worse | 0 | 0
  Data missing | 5 | 4

11. Secondary Outcome: Part A: Change From Baseline in Whole Body (WB) Longitudinal Composite Muscle Fat Infiltration (MFI) of B Muscles at Week 48
Description: The whole-body longitudinal composite muscle fat infiltration (MFI) of predefined B muscles is measured by musculoskeletal (MSK) magnetic resonance imaging (MRI). MFI quantifies the extent of fat replacement in muscle tissue, which is a key marker of disease progression in facioscapulohumeral muscular dystrophy (FSHD). The B muscles are a prespecified subset of muscles that are most relevant to FSHD progression. A decrease or smaller increase in MFI indicates slower disease progression or a potential treatment benefit. Change from Baseline was calculated as the post-treatment value minus the value at Baseline.
Time Frame: Baseline (Day 1) and at Week 48
Population: Full Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 114 | 113
Percent | 0.405 (0.893) | 0.551 (0.771)

12. Secondary Outcome: Part A: Relative Change From Baseline in Average Shoulder Abductor Strength by Hand-held Quantitative Dynamometry at Week 48
Description: Average shoulder abductor strength was assessed using hand-held dynamometry (HHD). Bilateral strength measurements were acquired from both upper limbs, with the average calculated for each participant. The relative change from baseline was expressed as a percentage. This evaluated the effect of losmapimod, relative to placebo, on muscle strength in individuals diagnosed with facioscapulohumeral muscular dystrophy (FSHD). Standardized procedures and equipment were employed across all study sites for strength testing, and trained personnel conducted all measurements to ensure consistency. Baseline is the last non-missing evaluation prior to first dose of study drug. Relative change from Baseline = 100 x (Post-baseline value - Baseline value) / (Baseline value).
Time Frame: Baseline (Day 1) and at Week 48
Population: Full Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 124 | 125
Percent | 17.38 (52.17) | 16.87 (56.81)

13. Secondary Outcome: Part A: Number of Participants Serious TEAEs and TEAEs
Description: as for outcome 2
Time Frame: Up to Week 48
Population: Safety Analysis Set comprises all participants who received any study drug in the placebo-controlled treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants
  Any non-serious TEAE | 122 | 112
  Any serious TEAE | 5 | 8

14. Secondary Outcome: Part A: Number of Participants With Clinically Significant Changes in Clinical Chemistry Parameters
Description: Blood samples were collected for the analysis of clinical chemistry parameters including Glucose, sodium, potassium, calcium, inorganic phosphate, total protein, albumin, blood urea nitrogen, creatinine, total bilirubin, direct bilirubin, alkaline phosphatase, aspartate aminotransferase, alanine aminotransferase, gamma-glutamyltransferase and creatine phosphokinase
Time Frame: Up to Week 48
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 0

15. Secondary Outcome: Part A: Number of Participants With Clinically Significant Changes in Hematology Parameters
Description: as for outcome 4
Time Frame: Up to Week 48
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 0

16. Secondary Outcome: Part A: Number of Participants With Clinically Significant Changes in Urinalysis
Description: as for outcome 5
Time Frame: Up to Week 48
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 0

17. Secondary Outcome: Part A: Number of Participants With Clinically Significant Changes in Vital Parameters
Description: as for outcome 6
Time Frame: Up to Week 48
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 0

18. Secondary Outcome: Part A: Number of Participants With Clinically Significant Changes in Electrocardiogram (ECG) Parameters
Description: Twelve-lead ECGs was performed after participants has been recumbent for at least 5 minutes.
Time Frame: Up to Week 48
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 0

19. Secondary Outcome: Part A: Number of Participants With Clinically Significant Changes in Physical Examinations
Description: as for outcome 8
Time Frame: Up to Week 48
Population: Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Losmapimod 15 Milligrams (mg) | Part A: Placebo
Number analyzed (Participants) | 130 | 130
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Part A: Up to 48 Weeks; Part B (OLE Period): Up to Week 127
Description: Serious TEAE and TEAE > 5% has been presented for Safety Analysis Set in Part A and Open-label Analysis Set in Part B. Safety Analysis Set comprises of all participants who received any study drug in the placebo-controlled treatment period. Open-Label Analysis Set comprises of all participants who received at least 1 dose of losmapimod in Part B.
Groups:
- Part A: Placebo-controlled Treatment Period: Losmapimod: Participants received Losmapimod 15 mg orally twice daily (BID) with food for 48 weeks.
- Part A: Placebo-controlled Treatment Period: Placebo: Participants received matching placebo orally twice daily (BID) with food for 48 weeks.
Arm/Group | Part A: Placebo-controlled Treatment Period: Losmapimod | Part A: Placebo-controlled Treatment Period: Placebo | Part B: Open Label Treatment Period: Losmapimod
All-Cause Mortality (participants affected / at risk) | 0/130 | 1/130 | 0/249
Serious Adverse Events (participants affected / at risk) | 5/130 | 8/130 | 7/249
Other Adverse Events (participants affected / at risk) | 122/130 | 112/130 | 94/249
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo-controlled Treatment Period: Losmapimod (N=130) | Part A: Placebo-controlled Treatment Period: Placebo (N=130) | Part B: Open Label Treatment Period: Losmapimod (N=249)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Peroneal nerve injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post ablation syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Placebo-controlled Treatment Period: Losmapimod (N=130) | Part A: Placebo-controlled Treatment Period: Placebo (N=130) | Part B: Open Label Treatment Period: Losmapimod (N=249)
COVID-19 (Infections and infestations) | 16 | 13 | 9
Influenza (Infections and infestations) | 6 | 8 | 5
Nasopharyngitis (Infections and infestations) | 30 | 29 | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 12 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 11 | 2
Diarrhoea (Gastrointestinal disorders) | 9 | 11 | 5
Nausea (Gastrointestinal disorders) | 7 | 7 | 4
Dizziness (Nervous system disorders) | 7 | 2 | 4
Headache (Nervous system disorders) | 16 | 16 | 11
Fall (Injury, poisoning and procedural complications) | 22 | 23 | 20
Rash (Skin and subcutaneous tissue disorders) | 7 | 1 | 3
Fatigue (General disorders) | 7 | 7 | 4
Influenza like illness (General disorders) | 8 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/70/NCT05397470/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT05397470/SAP_001.pdf